CLINICAL TRIAL: NCT07025564
Title: A Phase 1 Trial of miRisten in Adult Patients With Relapsed/Refractory AML
Brief Title: MiRisten for the Treatment of Relapsed or Refractory Acute Myeloid Leukemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24764; NCI-2025-03912 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24764 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2025-06-06; First posted 2025-06-17 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Recurrent Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Specimen Handling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (miRisten) (Experimental): Patients receive miRisten IV over 30 minutes BID on days 1-5, 8-12 and 15-19 in the absence of disease progression or unacceptable toxicity. Patients also undergo ECHO during screening and bone marrow and blood sample collection throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Echocardiography Test; Drug: miR-126 Inhibitor miRisten

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo bone marrow and blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Drug: miR-126 Inhibitor miRisten — Given IV
  Other Names: CpG-linked Anti-Mir-126 Oligonucleotide; miRisten; Oligodeoxynucleotide Anti-miR-126 Inhibitor miRisten; MicroRNA-126 Inhibitor miRisten; CpG(D19)-Anti-miR-126; ODN-based CpG-Anti-miRNA-126;

SUMMARY:
This phase I trial tests the safety, side effects, and best dose of miRisten in treating patients with acute myeloid leukemia (AML) that has come back after a period of improvement (relapsed) or that has not responded to previous treatment (refractory). MiRisten may stop the growth of cancer cells by blocking some of the molecules needed for cell growth. Giving miRisten may be safe, tolerable and/or effective in treating patients with relapsed or refractory AML.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the safety and tolerability of miR-126 inhibitor miRisten (miRisten) given intravenously (i.v.) twice daily.

II. Determine the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D).

SECONDARY OBJECTIVES:

I. Evaluate the anti-leukemic activity, as assessed by complete remission (complete response [CR]+complete response with Incomplete hematopoietic recovery [CRi]+CR with partial hematologic recovery [CRh]), overall response (overall response rate [ORR]: CR+CRi+CRh+partial response [PR]) and minimal residual disease negative (MRD-) rate and duration over the study period.

II. Estimate overall survival (OS), progression-free survival (PFS) and duration of response (DOR) rate at 6 months.

III. Describe the pharmacokinetics (PK) of miRisten.

EXPLORATORY STUDY OBJECTIVES:

I. Evaluate pharmacodynamics (PD) of miRisten therapy to identify biomarkers of clinical response and resistance.

II. Estimate miR-126 level in the bone marrow and blood pre-, post-therapy. III. Evaluate the impact of miRisten on miR-126 and its targets (e.g., SPRED1, CDK3, PIK3R2) in bone marrow.

IV. Estimate leukemia stem cell burden in bone marrow pre-, post-therapy. V. Monitor levels of cytokines and complement over time. VI. Dissect the mechanisms of miR-126-dependent leukemia stem cell (LSC) survival and self-renewal.

VII. Estimate the anti-leukemogenic force, therapeutic work induced by miRisten using the microRNA (miRNA)-based state transition model.

OUTLINE: This is a dose-escalation study.

Patients receive miRisten IV over 30 minutes twice a day (BID) on days 1-5, 8-12 and 15-19 in the absence of disease progression or unacceptable toxicity. Patients also undergo echocardiography (ECHO) during screening and bone marrow and blood sample collection throughout the trial.

After completion of study treatment, patients are followed up at 30 days and then at 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative.
* Agreement to allow the use of archival tissue from diagnostic tumor biopsies

  * If unavailable, exceptions may be granted with study principal investigator (PI) approval.
* ≥ 18 years.
* Eastern Cooperative Oncology Group (ECOG) ≤ 2.
* Patients with histologically confirmed AML, according to International Consensus Classification (ICC) or World Health Organization (WHO) criteria, with relapsed or refractory (R/R) disease who have failed treatment with, or are ineligible for, available therapies known to be active for treatment of AML.

  * Patients with extramedullary disease may be included if they also have concurrent marrow disease.
* Fully recovered from the acute toxic effects (except alopecia) to ≤ grade 1 to prior anti-cancer therapy.
* Life expectancy of ≥ 3 months.
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN) (performed within 28 days prior to day 1 of protocol therapy unless otherwise stated).
* Aspartate aminotransferase (AST) ≤ 3 x ULN (performed within 28 days prior to day 1 of protocol therapy unless otherwise stated).
* Alanine aminotransferase (ALT) ≤ 3 x ULN (performed within 28 days prior to day 1 of protocol therapy unless otherwise stated).
* Creatinine clearance of ≥ 60 mL/min per 24-hour urine test or the Cockcroft-Gault formula (performed within 28 days prior to day 1 of protocol therapy unless otherwise stated).
* International normalized ratio (INR) or prothrombin (PT) ≤ 1.5 x ULN (performed within 28 days prior to day 1 of protocol therapy unless otherwise stated).
* Activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN (performed within 28 days prior to day 1 of protocol therapy unless otherwise stated).
* Left ventricular ejection fraction (LVEF) ≥ 45% (performed within 28 days prior to day 1 of protocol therapy unless otherwise stated).
* Corrected QT interval (QTcF) ≤ 480 ms based on Fridericia's formula

  * Note: To be performed within 28 days prior to day 1 of protocol therapy.
* Women of childbearing potential (WOCBP): negative urine or serum pregnancy test (performed within 28 days prior to day 1 of protocol therapy unless otherwise stated).

  * If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Agreement by females and males of childbearing potential to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 3 months after the last dose of protocol therapy.

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only).

Exclusion Criteria:

* Allogeneic hematopoietic stem cell transplant within 3 months prior to day 1 of protocol therapy. Patients must be off calcineurin inhibitors for at least 2 weeks prior to day 1 of protocol therapy.
* Chemotherapy, radiation therapy, biological therapy, immunotherapy within 14 days prior to day 1 of protocol therapy, with the exception of hydroxyurea.
* Strong and moderate CYP3A4 inducers and strong CYP3A inhibitors (with the exception of azole antifungals) within 7 days prior to day 1 of protocol therapy.
* Foods/supplements that are strong inhibitors or strong or moderate inducers of CYP3A (such as St. John's wort) within 3 days prior to initiation of and during study treatment.
* Systemic steroid therapy > 10 mg/day (≤ 10mg/day prednisone equivalent ok) or any other form of immunosuppressive medication within 14 days. Inhaled or topical steroids, and adrenal replacement steroid doses ≤10 mg daily prednisone equivalent, are permitted. Steroids given for study drug infusion reaction prophylaxis or infusion reactions should not count towards this maximum.
* Must not have received or planning to receive live vaccine while being on study or 28 days before and after completion of treatment.
* Acute promyelocytic leukemia (APL).
* History of allergic or infusion reactions attributed to compounds of similar chemical or biologic composition to study agent.
* Inability to tolerate dexamethasone at the doses prescribed in this protocol.
* Unstable cardiac disease as defined by the following:

  * Unstable angina
  * Uncontrolled atrial fibrillation or hypertension
  * Acute coronary syndrome and/or revascularization (e.g., coronary artery bypass graft, stent) within 6 months of first dose of study drug.
* Clinically significant uncontrolled illness.
* Uncontrolled active infection.
* Other active malignancy. Patients with a prior or concurrent malignancy whose natural history or treatment have the potential to interfere with the safety or efficacy assessment of the investigational regimen are not eligible for this trial. Low grade indolent malignancies may be allowed if not actively undergoing treatment (such as non-melanoma skin cancers, low grade prostate cancer and others per the PI discretion).
* Females only: Pregnant or breastfeeding.
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures.
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-02-28 (Estimated); Primary Completion 2027-04-08 (Estimated); Study Completion 2027-04-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 30 days after completion of study treatment
  Toxicity data collection will include incidence and nature of adverse events (AEs) (including grade 3 and 4 AEs, treatment-related AEs, serious adverse events, dose limiting and moderate toxicities, AEs requiring discontinuation of miRisten, and changes in laboratory values.

SECONDARY OUTCOMES:
Disease response | Up to 6 months after completion of study treatment
  Will be assessed according to the European LeukemiaNet Criteria.
Duration of response | From the date of first documented response to documented disease relapse, progression or death whichever occurs first, assessed p to 6 months after completion of study treatment
  Will be estimated using the product-limit method of Kaplan and Meier.
Progression-free survival | From date of first dose of study drug to first documented evidence of disease progression or death from any cause, whichever occurs first, assessed up to 6 months after completion of study treatment
  Will be estimated using the product-limit method of Kaplan and Meier.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Blackmon, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States